CLINICAL TRIAL: NCT00002194
Title: An Open-Label Study in HIV+ Patients to Determine the Effects of Nevirapine (Viramune) on the Pharmacokinetics of Clarithromycin and Activity of Cytochrome 3A4.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 200G
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-08

CONDITIONS: HIV Infections
Keywords: Antibiotics, Macrolide; Clarithromycin; Nevirapine; Reverse Transcriptase Inhibitors; Cytochrome P-450; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Erythromycin; Nevirapine; Clarithromycin

INTERVENTIONS:
Drug: Erythromycin
Drug: Nevirapine
Drug: Clarithromycin

SUMMARY:
To evaluate the potential pharmacokinetic interaction between nevirapine and clarithromycin, and to determine the effects of nevirapine on cytochrome P450 3A4 (CYP3A4) activity in vivo.

DETAILED DESCRIPTION:
The study is conducted in two separate groups. Patients in Group I receive clarithromycin orally for 32 days and nevirapine orally for 28 days.

Patients in Group II receive erythromycin intravenously on days 0, 14, 28, and 43 and nevirapine orally for 28 days.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

Antiretroviral drugs (i.e., zidovudine, zalcitabine, stavudine, lamivudine, didanosine, indinavir, saquinavir) provided that there has been no change in dosing of the medication > 25% within 4 weeks of study entry.

Patients must have:

* HIV positive status.
* CD4 count >= 100 cells/mm3.

Prior Medication:

Allowed:

Patients may be on clarithromycin at study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions are excluded:

Malabsorption, severe chronic diarrhea, or inability to maintain adequate oral intake.

Concurrent Medication:

Excluded:

Macrolide antibiotics (erythromycin, azithromycin, dirithromycin), azole fungals (ketoconazole, fluconazole, itraconazole), rifampin, rifabutin, phenytoin, terfenadine, astemizole, cisapride, triazolam, midazolam, other non-nucleoside reverse transcriptase inhibitors, antibiotics containing clavulanic acid, and Augmentin.

Patients with the following prior conditions are excluded:

* History of drug allergy or known drug hypersensitivity.
* History of clinically important disease including hepatic, renal, cardiovascular, or gastrointestinal disease.

Prior Medication:

Excluded:

* Investigational drugs or antineoplastic agents within 12 weeks of study entry.
* Participation in a clinical trial that used ERMBY within one year of study entry.
* Systemic treatment with drugs known to be potent hepatic enzyme inducers or inhibitors (e.g., oral macrolide antibiotics, azole antifungals, cimetidine, rifampin, rifabutin, and carbamazepine) within 28 days of study entry.
* Use of protease inhibitors; ritonavir, nelfinavir, indinavir, or non-nucleoside reverse transcriptase inhibitor compounds e.g., delavirdine) within 4 weeks of study entry.

Prior Treatment:

Excluded:

Radiotherapy within 12 weeks of study entry.

Risk Behavior:

Excluded:

Current history (within the last year) of IVDA, ETOH, or substance abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36

CONTACTS AND LOCATIONS:
Locations (1):
- South Florida Bioavailability Clinic, Miami, Florida, United States